CLINICAL TRIAL: NCT05068375
Title: Unusual Pattern of Thrombotic Events in Young Adults Noncritically Ill Patients With COVID-19 May Result From An Un-diagnosed Inherited Form of Thrombophilia
Brief Title: Unleash the Mystery of COVID-19 Related Unusual Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Ibrahim Yousef, Assistant Professor MD Phd., Sohag University
Other Study IDs: Soh-Med-21-04-39
Record Dates: First submitted 2021-10-02; First posted 2021-10-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thrombotic group: Non-critically COVID-19 patients with unusual thrombotic events
  Interventions: Diagnostic Test: Thrombophilia screening
- Non-thrombotic group: Non-critically COVID-19 patients without thrombotic events

INTERVENTIONS:
Diagnostic Test: Thrombophilia screening — Genetic thrombophilia and acquired thrombophilia screening
  Groups: Thrombotic group

SUMMARY:
Arterial thrombosis and unusual patterns of thrombotic events in young adults patients with COVID-19 are yet rarely described in this setting and could be underestimated. There is a real need for studies to describe the frequency of unusual thrombotic complications.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), first identified in Wuhan, China in December of 2019, has become a worldwide pandemic with widespread illness and mortality. Clinical manifestations of Coronavirus disease 2019 (COVID-19) are absent or mild in a substantial proportion of patients who test positive for COVID-19. Although respiratory compromise is the cardinal feature of the disease, early studies have suggested that elevated circulating D-dimer levels are associated with mortality suggesting a distinct coagulation disorder associated with COVID-19. COVID-19 infection is commonly complicated with pro-thrombotic state and endothelial dysfunction.

Recent autopsy studies of COVID-19 patients supported this hypothesis by demonstrating the extensive extracellular fibrin deposition and presence of fibrin thrombi within distended capillaries and small vessels. Observational studies reported an excess of venous thromboembolic events (deep vein thrombosis (DVT), pulmonary embolism (PE)) among patients suffering from Covid-19. Retrospective studies have reported thrombotic rates in excess of 20% to 30%, but the use of prophylactic anticoagulation and duration of treatment were not consistent between studies. Unrecognized PE and pulmonary in situ thrombosis were reported as causes of the high mortality observed among COVID-19 patients. There is currently no clear estimation of the risk of arterial and, in particular, venous thromboembolic complications which depend on local diagnostic and pharmacological preventive strategies. In addition to D-dimer, a prolonged prothrombin time (PT) has been associated with decreased survival and increased need for critical care.

However, arterial thrombosis and unusual patterns of thrombotic events in young adults patients with COVID-19 are yet rarely described in this setting and could be underestimated (9). Thus, there is a real need for studies to describe the frequency of unusual thrombotic complications. Therefore, the purpose of this study will be to explore thromboembolic risk and associated predicting factors in the young adults' cohort of noncritically ill COVID-19 patients which will help to optimize diagnostic, therapeutic, and preventive strategies of COVID-19 related thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* non-critically ill young adults' patients with COVID-19 admitted to our hospital will have confirmed unusual thrombotic events and accept recruitment to this study.

After that, we will focus only on previously healthy patients without pre-existing prothrombotic factors and presented with COVID-19 related unusual thrombotic events

Exclusion Criteria:

* COVID-19 patients below 18 years and above 40 years
* COVID-19 patients diagnosed as critically ill COVID-19
* COVID-19 patients with pre-existing diabetes mellitus (DM), hypertension, ischemic heart disease (IHD), valvular heart disease, cardiomyopathy and chronic arrhythmia, dyslipidemia, metabolic syndrome, chronic kidney disease, liver disease, nephrotic syndrome, previous autoimmune disease, and malignancy
* COVID-19 patients with chronic lung disease or immune compromise
* COVID-19 pregnant women
* COVID-19 patient with history of thrombosis/ psychiatric disorders/ drug abuse
* COVID-19 patient previously diagnosis with congenital thrombophilia
* COVID-19 patient with drug history could induce thrombosis.
* COVID-19 patient unwilling to be followed up.

  * Patients are previously diagnosed with one or more risk factors of thrombosis

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: - Study group:
  At Sohag University Hospitals, we conducted a longitudinal observational study with a 6-month follow-up duration across a fourteen-month period (April 2020 to June 2021). This study enrolled young adult non-critical ill patients (age 18 to 40) with a positive SARS-CoV-2 reverse-transcriptase polymerase chain reaction (rt-PCR) test and unusual sites of thrombotic events. These patients will be compared to young adult non-critical patients presented to our hospital with COVID-19 without thrombosis during the study period.
  Patients will be classified into two groups:
  * Group I: COVID-19 patients with unusual thrombosis
  * Group II: COVID-19 patients without unusual thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Frequency | Form April 2020 to April 2021
  Rates of unusual thrombotic events among non-critically ill young adults' patients with COVID-19
Thrombosis progression | First month after diagnosis
  Thrombosis progression: Symptomatic extension of a pre-existing thrombus or new symptomatic thrombus not evident on the initial imaging at a second compressive examination.
Bleeding complications of the UTEs | First month after diagnosis
  Bleeding (major, minor bleedings)
  I. Major bleeding is defined as frank bleeding contributed to death or associated with a decreasing in hemoglobin ≥2 g/dL, or need a packed red blood cells transfusion ≥2 units, or bleeding at a critical site.
  II. Non-major bleeding was defined as any symptom or sign of bleeding that did not fit the criteria of major bleeding but fulfilled at least one of the these criteria: leading to hospitalization, or requiring healthcare professional medical intervention, or spurring a face-to-face assessment.
Mortality | First month after diagnosis
  Death frequency

SECONDARY OUTCOMES:
Thrombosis recurrence | During 6 months of follow up period
  Incidence of thrombosis recurrence after the initial thrombotic event(s)
Bleeding | During 6 months of follow up period
  Incidence of bleeding (major, minor bleedings)
Mortality | During 6 months of follow up period
  Death frequency

CONTACTS AND LOCATIONS:
Locations (1):
- , Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No